CLINICAL TRIAL: NCT00654251
Title: Utility Of Home Based Gait Monitoring, Performance Scores And Functional Visual Assessment In Spinocerebellar Ataxias (SCA)
Brief Title: Measuring Neurological Impairment and Functional Visual Assessment In Spinocerebellar Ataxias
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of Texas (Other)
Responsible Party: James J Corbett, University of Mississippi Medical Center
Other Study IDs: 2007-0228
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Spinocerebellar Ataxia
Keywords: Spinocerebellar ataxia; Machado-Joseph disease; Gait monitoring; Functional vision assessment
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Measuring the various difficulties patients with spinocerebellar ataxias (SCA) report in an accurate manner is important to be able to test any therapy that may be developed. As basic research identifies some therapy of this type, clinicians are planning studies that can either prove or disprove that such treatments actually have an effect. Walking problems and problems with eye movements that can give rise to visual complaints are common in the SCA's.

Existing neurological scales such as the "SARA" are based on the usual neurological examination items that can carry a degree of subjective bias. Also the intervals between numbers on such scores often do not carry the same "weight" so that the difference between a score of 1 and 2 may not be equal to difference between 2 and 3. Lastly, such scales done in the clinic setting capture only a brief period of a patient's day. We propose that examination of home based gait monitoring, timed tests of motor function and quantitative measures of visual problems in patients with SCA are more useful in measuring the disability in these patients.

DETAILED DESCRIPTION:
Spinocerebellar ataxias (SCA's) are relatively rare, inherited disorders of the cerebellum that cause inexorably progressive imbalance and incoordination as well as speech problems. Recent molecular genetic studies have raised hopes for meaningful treatments for these conditions. Before one can embark on therapeutic studies on the SCA's it is essential that we have validated instruments for measuring disease progression. Rating scales based on neurological examinations have been reported recently but their sensitivity to change and reproducibility are still being examined. In an attempt to produce readily quantifiable and sensitive measures of motor function in the SCA's, we are proposing to examine the utility of home based gait monitoring, timed tests of motor function and quantitative measures of visual problems in patients with SCA's. These measurements which will produce continuous rather than categorical variables, and may be subject to less arbitrariness on the part of the examiner, are hypothesized to be not only valid measures but also more sensitive.

The overall aim of the project is to assess the utility of home based gait monitoring, timed performance measures and functional visual testing as measures to monitor disease progression in SCA's. The concurrent validity of these measures will be tested by correlating them with an established examination based ataxia scale (Scale for assessment and rating of ataxia: SARA), an activity of daily living scale (Barthel index) and functional staging.

Aim 1: Hypothesis: Motor impairment in SCA's can be assessed validly in the home setting by utilizing the step activity monitor (SAM).

Aim 2: Hypothesis: Motor impairment in SCA's can be further quantified using performance measures: the 9-hole peg board test and the timed 25 foot walk.

Aim 3: Hypothesis: Visual problems reported by patients with SCA's can be quantified by low contrast vision testing, stereoacuity measures, color vision and vergence amplitudes utilizing well-established ophthalmologic techniques.

Aim 4: Hypothesis: The neurological impairment as measured by these measures will correlate with each other, with scores on SARA, with the Barthel index score and with functional staging.

Aim 5: Hypothesis: Ataxia grading using the SAM, timed performance measures and functional visual scores will be more sensitive than SARA for measuring disease progression

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of Spinocerebellar Ataxia (Type 1,2,3,6,7,8 and 10) will be selected from those attending the ataxia clinic in the Neurology Department at University of Mississippi Medical Center
2. Patients will be 18years or older in age
3. All patients are able to walk with or without assisted devices

Exclusion Criteria:

1. Patients less than 18years.
2. Patients who are wheelchair bound

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Ataxia Clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Home based gait data vs SARA index | 0, 6, 12, 24 months

SECONDARY OUTCOMES:
Barthel Index | 0, 6, 12, 24 months
Visual function- acuity, contrast, stereo, color | 0, 6, 12, 24 months
Ocular Motility defects- phoria/tropia, vergence amplitudes | 0, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James J Corbett, MD, Study Chair — University of Mississippi Medical Center; S H Subramony, MD, Study Director — University of Texas; Sachin Kedar, MD, Study Director — University of Mississippi Medical Center
Locations (2):
- United States (2):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Texas Medical Branch, Galveston, Texas

REFERENCES:
- [Background] Schols L, Bauer P, Schmidt T, Schulte T, Riess O. Autosomal dominant cerebellar ataxias: clinical features, genetics, and pathogenesis. Lancet Neurol. 2004 May;3(5):291-304. doi: 10.1016/S1474-4422(04)00737-9. PMID 15099544
- [Background] Duenas AM, Goold R, Giunti P. Molecular pathogenesis of spinocerebellar ataxias. Brain. 2006 Jun;129(Pt 6):1357-70. doi: 10.1093/brain/awl081. Epub 2006 Apr 13. PMID 16613893
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946
- [Background] Subramony SH, May W, Lynch D, Gomez C, Fischbeck K, Hallett M, Taylor P, Wilson R, Ashizawa T; Cooperative Ataxia Group. Measuring Friedreich ataxia: Interrater reliability of a neurologic rating scale. Neurology. 2005 Apr 12;64(7):1261-2. doi: 10.1212/01.WNL.0000156802.15466.79. PMID 15824358
- [Background] Busse ME, Pearson OR, Van Deursen R, Wiles CM. Quantified measurement of activity provides insight into motor function and recovery in neurological disease. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):884-8. doi: 10.1136/jnnp.2003.020180. PMID 15146006
- [Background] Fahey MC, Corben LA, Collins V, Churchyard AJ, Delatycki MB. The 25-foot walk velocity accurately measures real world ambulation in Friedreich ataxia. Neurology. 2007 Feb 27;68(9):705-6. doi: 10.1212/01.wnl.0000256037.63832.6f. No abstract available. PMID 17325285